CLINICAL TRIAL: NCT05734898
Title: NKG2D CAR-NK Cell Therapy for the Treatment of Patients With Relapsed and/or Refractory Acute Myeloid Leukemia
Brief Title: NKG2D CAR-NK & r/rAML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Cheetah Cell Therapeutics Co., Ltd (Other)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2023]TXB--001
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: AML
Keywords: CAR-NK; NKG2D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rrAML (Experimental)
  Interventions: Biological: NKG2D CAR-NK

INTERVENTIONS:
Biological: NKG2D CAR-NK — Lymphodepleting chemotherapy followed by NKG2D CAR-NK infusion

SUMMARY:
This trial will explore the maximum tolerated dose（MTD）of NKG2D CAR-NK cells in the treatment of relapsed or/and refractory AML in a dose-escalation manner, and observe the clinical safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 3 years old and ≤ 75 years old, male or female;
2. Meet the diagnostic criteria for recurrent AML specified in the guidelines for diagnosis and treatment of acute myelogenous leukemia (relapse/refractory) in China (2017): leukemic cells reappear in peripheral blood or bone marrow MRD > 0.1% after complete remission (CR), including relapse after allogeneic hematopoietic stem cell transplantation or extramedullary leukemic cell infiltration.
3. Meet the diagnostic criteria for refractory AML specified in the guidelines for diagnosis and treatment of acute myelogenous leukemia (relapse/refractory) in China (2017): Initial cases with failure of 2 lines of standard treatment; patients who relapsed within 12 months after consolidation intensification after CR; recurrence in 12 months and no respond to conventional chemotherapy; 2 or more recurrences; persistent extramedullarial leukemia;
4. Patients currently have no effective treatment options, such as chemotherapy or allogeneic hematopoietic stem cell transplantation, or patients voluntarily choose to infuse NKG2D CAR-NK cells as the first treatment option;
5. Physical status assessment (ECOG-PS) of the Eastern Oncology Collaborative Group is 0-2 points;
6. Life expectancy ≥ 12 weeks from the time of enrollment;
7. The main organs of the patient are well functioned: (1) cardiac function: no heart disease or coronary heart disease, the patient's cardiac function grade 1-2; (2) liver function: TBIL≦3ULN, AST≦2.5ULN, ALT≦2.5ULN; (3) Renal function: Cr≦1.25ULN;
8. Flow cytometry check for NKG2D ligand expression on the surface of cancer cells as a reference for patient selection;
9. The patient's peripheral superficial vein is accessible for IV insertion and blood draws;
10. No other serious diseases that conflict with this protocol (e.g., autoimmune diseases, immunodeficiency, organ transplantation);
11. No history of other malignant tumors;12. Women of childbearing age must be tested negative for pregnancy within 7 days, and subjects of childbearing age must use appropriate contraception during both the trial and for 3 months after the test;

13. Subjects have negative HIV, HBV, HCV, syphilis serology test results; 14. Written informed consent form must be signed by the patient or the patient's immediate family members before enrollment.

Exclusion Criteria:

1. Acute promyelocytic leukemia (Type M3);
2. Patients with cardiac insufficiency, patients with liver and renal insufficiency;
3. Patients with other malignant tumors need to be treated;
4. Poorly controlled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >90 mmHg) or clinically significant cardiovascular and cerebrovascular diseases such as cerebrovascular accident (within 6 months before signing the informed consent form), myocardial infarction (within 6 months before signing the informed consent), unstable angina, congestive heart failure, or severe arrhythmias that cannot be controlled with drugs or have a potential impact on research treatment;
5. Patients suffering from other hematologic diseases (such as hemophilia, myelofibrosis, etc., which researchers consider unsuitable for enrollment);
6. Patients with diffuse vascular internal coagulation;
7. Patients with concomitant serious infection or other serious underlying medical condition;
8. Patients with variable immunodeficiency and autoimmune diseases;
9. Patients who have severe allergic diseases;
10. Clinical symptoms of brain dysfunction or severe mental illness that can not understand or follow the research protocol;
11. Have participated in clinical trials of other drugs within 4 weeks or within 21 days of surgery;
12. Have received cell therapy in the previous 1 month;
13. Have received hormonal drug therapy in the previous 14 days;
14. Known human immunodeficiency virus (HIV) seropositivity or active hepatitis B or C infection or syphilis;
15. Have received organ transplants (excluding stem cell transplant patients);
16. Drug abuse, medical, psychological or social conditions that may interfere with a subject's participation in the study or evaluation of the results of the study;
17. Pregnant or lactating women;
18. Those who cannot be followed up as scheduled;
19. Patients, who in the opinion of the investigator, have any clinical or laboratory abnormalities or compliance problems and are not suitable to participate in this clinical study.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days
  Dose-Limiting Toxicity
MTD | 28 days
  Maximal Tolerable Dose

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No